CLINICAL TRIAL: NCT02054559
Title: Randomized Phase III Trial Comparing R-CHOP Alone and R-CHOP Plus Radiotherapy for Localized CD20+ Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: R-CHOP Alone vs. R-CHOP Plus Radiotherapy for Localized CD20+ DLBCL
Acronym: ASPIRE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No consensus among trial centers regarding protocol
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Cheolwon Suh, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC_NHL02
Record Dates: First submitted 2014-01-29; First posted 2014-02-04 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: localized; diffuse large B-cell lymphoma; R-CHOP chemotherapy; radiotherapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — R-CHOP protocol; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Total 6 cycles of R-CHOP (Active Comparator)
  Interventions: Drug: R-CHOP
- Total 3 cycles of R-CHOP + RT (Experimental): Total 3 cycles of R-CHOP followed by radiotherapy (involved field or involved site radiotherapy, 30-50 Gy/ 15-25 fractions)
  Interventions: Drug: R-CHOP; Radiation: Radiotherapy

INTERVENTIONS:
Drug: R-CHOP — R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, prednisone (or prednisolone))
Radiation: Radiotherapy
  Arms: Total 3 cycles of R-CHOP + RT

SUMMARY:
To compare the efficacy and safety of chemotherapy alone and combined modality therapy in the treatment of localized CD20 (+) diffuse large B-cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Histologically confirmed CD20-positive Diffuse Large B-cell Lymphoma (DLBCL), NOS
* Immunostains for CD20, CD5, CD3, CD10, MUM-1, BCL-6, BCL-2 and Ki-67 and the in situ hybridization for Epstein-Barr virus are recommended for diagnosis of DLBCL, NOS.
* No prior treatment for DLBCL
* Stage I or contiguous II disease (Involvement of two adjacent lymph node regions or organ involvement with regional lymph nodes)
* Performance status: ECOG 0-2.
* Age ≥ 18 years
* Cardiac ejection fraction ≥ 45% as measured by MUGA or 2D ECHO without clinically significant abnormalities
* Adequate renal function: serum creatinine level < 2 mg/dL
* Adequate liver functions
* Adequate hematological function: hemoglobin ≥ 9.0 g/dL absolute neutrophil count (ANC) ≥ 1,500/μL and platelet count ≥ 75,000/μL, unless abnormalities are due to bone marrow involvement by lymphoma
* Life expectancy >= 6 months
* A negative serum or urine pregnancy test prior to treatment must be available both for pre menopausal women and for women who are < 1 years after the onset of menopause.
* Female patients of child bearing potential must use an effective method of birth control (i.e. hormonal contraceptive, intrauterine device,diaphragm with spermicide, condom with spermicide or abstinence) during treatment period and 1 month thereafter; Males must use an effective method of birth control during treatment period and 3 months thereafter.

Exclusion Criteria:

* Other subtypes NHL than CD20 (+) DLBCL, NOS
* Transformed DLBCL from follicular lymphoma or other indolent lymphomas
* Bulky disease ( longest diameter >=10 cm)
* Previous treatment for DLBCL with immunotherapy or chemotherapy except for short-term corticosteroids (duration of ≤ 8 days) before inclusion
* CNS involvement by lymphoma or any evidence of spinal cord compression.
* Primary Central Nervous System (CNS) DLBCL
* Primary testicular lymphoma
* Primary breast lymphoma
* Patients with a known history of HIV seropositivity or HCV (+). (Patients who have HBV (+) are eligible. However, primary prophylaxis using antiviral agents (i.e. lamivudine, etc) is recommended for HBV carrier to prevent HBV reactivation during whole treatment period.)
* Prior history of malignancies other than lymphoma (except for basal cell or squamous cell carcinoma of the skin, early gastric cancer or carcinoma in situ of the cervix or breast or untreated prostatic cancer without any plan for a treatment) unless the patient has been free of the disease for ≥ 3 years
* Pregnant or lactating women
* Men who are not surgically sterile and women of childbearing potential not employing adequate contraception
* Other serious illness or medical conditions
* Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry
* History of significant neurological or psychiatric disorders including dementia or seizures
* Active uncontrolled infection (viral, bacterial or fungal infection)
* Other serious medical illnesses
* Known hypersensitivity to any of the study drugs or its ingredients
* Concomitant administration of any other experimental drug under investigation, or concomitant chemotherapy, hormonal therapy, or immunotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
To compare 3-year event-free survival | 3 years
  definition of events: failure to achieve CR after completion of planned 1st-line treatment, progression of disease, relapse, institution of a new anticancer treatment or any cause of death) rate in patients with CD20 (+) diffuse large B-cell lymphoma treated with either R-CHOP chemotherapy alone or R-CHOP plus radiotherapy

SECONDARY OUTCOMES:
To evaluate and compare OS between the two arms | 3 years
To evaluate and compare the ORR and CR rate | after completion of treatment
To evaluate and compare disease-free survival (DFS) | 3 years
To evaluate treatment-failure pattern | 3 years
Number of Participants with Adverse Events in each arm | 3 years
To assess patient-reported outcomes (PROs) in both arms | 3 years
A role of interim PET after 3 cycles of R-CHOP chemotherapy: correlation with PFS and OS | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea